CLINICAL TRIAL: NCT04629365
Title: Effects of Two Months of Ketogenic Diet on Body Composition, Muscle Strength and Blood Parameters in Competitive Natural Body Builders
Brief Title: Effects of Ketogenic Diet in Body Builders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Antonio Paoli, Full Professor, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BBKeto
Record Dates: First submitted 2020-11-09; First posted 2020-11-16 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Diet, Healthy; Body Weight
Keywords: ketogenic diet; body builders; athletes; body composition; hormones
MeSH Terms: conditions — Body Weight | interventions — Diet, Ketogenic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor treated anonymus data
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic Diet (Experimental): KD group consumed less than 50g/day of carbohydrates
  Interventions: Other: Ketogenic Diet
- Normal Diet (Active Comparator): ND group consumed 55% of the caloric intake from carbohydrates
  Interventions: Other: Normal Diet

INTERVENTIONS:
Other: Ketogenic Diet — KD group consumed less than 50g/day of carbohydrates
  Arms: Ketogenic Diet
Other: Normal Diet — ND group consumed 55% of the caloric intake from carbohydrates
  Arms: Normal Diet

SUMMARY:
the study sought to investigate the influence of 8 weeks of a very low carbohydrate ketogenic diet on body composition, muscle strength, muscle area and blood parameters in competitive natural body builders.

DETAILED DESCRIPTION:
nineteen natural body builders were randomly assigned to a ketogenic diet (KD) group or to a normal diet group (ND) with a traditional meal pattern. The two diets were isocaloric and included the same amount of protein per kg of body weight; but differed in the distribution of fats and carbohydrates; the latter were kept below 5% daily (less than 50g/day) in the KD group while represented 55% of the caloric intake in the WD group During the experimental period, training loads were similar in the two groups. Athletes were tested before and after 8 weeks of the intervention. Body composition , basal metabolism, muscle strength and blood parameters were measured.

ELIGIBILITY:
Inclusion Criteria:

* at least 5 years of training experiences
* competing in recognized body building category

Exclusion Criteria:

* adherence to special diets
* use of nutritional supplements (except a daily multivitamin-mineral and/or protein supplement)
* use of medications (steroids)
* diabetes or metabolic diseases

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Fat Mass | 8 weeks
  fat mass measured through body impedence analyser
Lean Body Mass | 8 weeks
  lean body mass mass measured through body impedence analyser
Maximal muscle strength | 8 weeks
  muscle strength measured via 1-RM test

SECONDARY OUTCOMES:
blood glucose | 8 weeks
  glucose as milligram per deciliter
testosterone | 8 weeks
  Testosterone free as picogram per milliliter
inflammatory cytokines | 8 weeks
  IL6, IL1β, TNFα measured as nanogram per deciliter
resting metabolism | 8 weeks
  resting energy expenditure measured as Kcal / day

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Paoli, MD, Principal Investigator — University of Padova
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy